CLINICAL TRIAL: NCT06688630
Title: The Effect of Laser Acupuncture on the Signs and Symptoms of Dry Eye Disease Due to Visual Display Terminal Use
Brief Title: Laser Acupuncture for Dry Eye Disease Due to Visual Display Terminal Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Inria Chandra, Resident of Medical Acupuncture Study Program, Indonesia University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 24-09-1470
Record Dates: First submitted 2024-11-12; First posted 2024-11-14 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: This study will compare the combination of laser acupuncture therapy and artificial tears with the combination of sham laser acupuncture therapy and artificial tears.
  The laser acupuncture and artificial tears therapy will be designated as the intervention group, while the sham laser acupuncture and artificial tears therapy will be designated as the control group.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participants, the ophthalmologist conducting the eye examinations, and the outcome assessors will be blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The laser acupuncture and artificial tears therapy
  Interventions: Device: The laser acupuncture and artificial tears therapy
- Control Group (Sham Comparator): The sham laser acupuncture and artificial tears therapy
  Interventions: Device: The sham laser acupuncture and artificial tears therapy

INTERVENTIONS:
Device: The laser acupuncture and artificial tears therapy — Laser acupuncture therapy is the application of a Reimers & Janssen LaserPen, with a power of 150mW and a wavelength of 810nm, alternating between Nogier frequencies A and C. The dosage is 2 joules per point, with a therapy duration of 26 seconds per point, targeting bilateral acupuncture points BL2, TE23, ST2, LI4, and ST36. The LaserPen is applied without pressing the laser probe onto the body surface.
  Artificial tears containing carboxymethylcellulose (CMC) will be used. The frequency of application is four times daily (morning, afternoon, evening, and night), with one drop per eye, administered to both eyes. Artificial tears will be used throughout the study duration (4 weeks). Use of any artificial tears other than CMC will be discontinued for 3 days and resumed on day 4 with CMC.
  Arms: Intervention Group
Device: The sham laser acupuncture and artificial tears therapy — Laser acupuncture therapy is a procedure using the same device but without activating the laser, so no energy is emitted. Performed at the same points as laser acupuncture therapy.
  Artificial tears containing carboxymethylcellulose (CMC) will be used. The frequency of application is four times daily (morning, afternoon, evening, and night), with one drop per eye, administered to both eyes. Artificial tears will be used throughout the study duration (4 weeks). Use of any artificial tears other than CMC will be discontinued for 3 days and resumed on day 4 with CMC.
  Arms: Control Group

SUMMARY:
The purpose of this clinical trial is to determine whether laser acupuncture can alleviate dry eye symptoms caused by visual display terminal use and to assess the safety of laser acupuncture. The research questions to be addressed are:

* Can laser acupuncture and artificial tears reduce the Ocular Surface Disease Index (OSDI) score, Tear Break-Up Time (TBUT) score, Ocular Surface Staining (OSS) score, and Schirmer Test score?
* Are there any side effects associated with laser acupuncture therapy?

The researchers will compare laser acupuncture and artificial tears with sham laser acupuncture (a procedure using the same device but without activating the laser, so no energy is emitted) to assess whether laser acupuncture and artificial tears can effectively treat dry eye associated with visual display terminal use.

Participants will:

* Receive either laser acupuncture therapy or sham laser acupuncture therapy for 6 sessions, twice a week, over a 3-week period.
* Use artificial tears daily, 4 times per day (morning, afternoon, evening, and night), with one drop per eye for both eyes, over a 4-week period.
* Attend follow-up visits at the eye clinic at baseline (before therapy), in week 2, and in week 4.
* Record any side effects observed after each session of laser acupuncture therapy.

DETAILED DESCRIPTION:
* Dry eye disease is an ocular condition characterized by common symptoms such as eye irritation, a sensation of grittiness, foreign body sensation, stickiness, itchiness, eye fatigue, redness, stabbing or burning sensations, increased blinking frequency, and symptom exacerbation in the afternoon or evening.
* Visual Display Terminal (VDT) refers to devices equipped with a screen for displaying graphics or digital content for specific tasks, commonly known as gadgets. Examples of VDTs include computers, laptops, televisions, and mobile phones.
* The Ocular Surface Disease Index (OSDI) is a questionnaire consisting of 12 questions designed to assess symptoms of dry eye, visual function, and environmental factors that may trigger dry eye.
* The Visual Analog Scale (VAS) is a scoring tool to measure the intensity of discomfort associated with dry eye, using a scale from 0 to 100, where 0 indicates "no pain/discomfort" and 100 indicates "the most severe pain/discomfort."
* Tear Break-Up Time (TBUT) is an examination used to assess how long the tear film remains on the ocular surface after blinking, as a measure for diagnosing dry eye. This test is conducted by an ophthalmologist.
* Ocular Surface Staining (OSS) is an examination in which dye is applied to the ocular surface to detect abnormalities on the eye's surface. This test is also performed by an ophthalmologist.
* The Schirmer test is a quantitative test used to measure tear volume over a period of 5 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18 - 59 years with dry eye complaints
* Diagnosed with DED by an Ophthalmologist with the criteria OSDI value ≥ 13, and TBUT value < 10 seconds
* Using VDT for at least 4 hours a day
* Not currently receiving other DED therapy other than CMC artificial tears
* Willing to participate in the study until completion and sign the informed consent

Exclusion Criteria:

* Acute infection or trauma to the eye and periorbita
* Eyelid abnormalities or facial paresis that prevent the eye from closing
* History of intraocular or extraocular surgery within the last 12 months
* Previously diagnosed with Steven Johnson Syndrome, Sjogren Syndrome, or diabetes mellitus
* Undergoing chemotherapy or post-chemotherapy
* Pregnant and lactating women
* Menopausal women or those receiving hormone therapy
* History of uncontrolled seizures or epilepsy

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2024-12-27 (Actual); Primary Completion 2025-03-14 (Actual); Study Completion 2025-03-14 (Actual)

PRIMARY OUTCOMES:
The Ocular Surface Disease Index | Before therapy, week 2, week 4
  The Ocular Surface Disease Index (OSDI) is a questionnaire consisting of 12 questions designed to assess symptoms of dry eye, visual function, and environmental factors that may trigger dry eye.
The Tear Break-up Time | Before therapy, week 2, week 4
  Tear Break-Up Time (TBUT) is an examination used to assess how long the tear film remains on the ocular surface after blinking, as a measure for diagnosing dry eye. This test is conducted by an ophthalmologist.

SECONDARY OUTCOMES:
The Ocular Surface Staining Score | Before therapy, week 2, week 4
  Ocular Surface Staining (OSS) score is a scoring of examination in which dye is applied to the ocular surface to detect abnormalities on the eye's surface.
The Schirmer Score | Before therapy, week 2, week 4
  The Schirmer score is an accumulation of tear volume over a period of 5 minutes.
The Visual Analog Scale | Before therapy, week 2, week 4
  The Visual Analog Scale (VAS) is a scoring tool to measure the intensity of discomfort associated with dry eye, using a scale from 0 to 100, where 0 indicates "no pain/discomfort" and 100 indicates "the most severe pain/discomfort."
Adverse Event | Up to week 4
  Symptoms reported by patients after receiving laser acupuncture therapy.

CONTACTS AND LOCATIONS:
Overall Officials: KPEK FKUI-RSCM, Principal Investigator — The Health Research Ethics Commitee ofFaculty of Medicine Universitas Indonesia - RSCM
Locations (1):
- Universitas Indonesia, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No